CLINICAL TRIAL: NCT06318728
Title: Musculotendinous Adaptations Induced by Training and Competitions in High and Low-performance Triathletes
Brief Title: Musculotendinous Adaptations in High and Low- Performance Triathletes
Acronym: MAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Sponsor
Other Study IDs: CAEE - 70162723.0.0000.8093
Record Dates: First submitted 2024-01-10; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2023-11

CONDITIONS: Athletes
Keywords: Triathlon; Achilles tendon; Triceps sural; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High Performance Triathletes Groups: Triathletes who have been practicing the sport for more than 2 years, can maintain a running pace in triathlon competition below 4 minutes and 10 seconds per kilometer for men and 4 minutes and 30 seconds per kilometer for women, and have a weekly running volume exceeding 35 kilometers.
- Low Performance Triathletes Groups: Triathletes who have completed at least 2 races, maintain a running pace in triathlon competition above 4 minutes and 50 seconds per kilometer for men and 5 minutes and 10 seconds per kilometer for women, and have a weekly running volume below 30 kilometers.
- Control Group: Physically active individuals, aged between 17 and 52 years, who do not engage in regular running.

SUMMARY:
This study aims to investigate the musculotendinous adaptations in the Achilles tendon and the muscles composing the triceps surae induced by triathlon training and competitions in high-performance and low-performance athletes. Twenty high-performance triathletes, twenty low-performance triathletes, and twenty physically active and healthy individuals of both genders will be recruited to constitute the research groups. Ultrasonography will be employed as the assessment method for the structures of the Achilles tendon and the muscular architecture of the triceps surae. The quality and portability of ultrasonography, coupled with its real-time information capabilities, make it the appropriate choice for this evaluation. The VISA-A scale (Victorian Institute of Sport Achilles Assessment) will be used to measure pain and function of the Achilles tendon. The reliability of ultrasonography measures will be obtained by evaluating images of individuals using the intraclass correlation coefficient, allowing for the analysis of result reproducibility. Data analysis will involve comparisons among the high-performance, low-performance, and physically active groups, aiming to identify differences in musculotendinous adaptations related to performance and injury predisposition. Structural changes occurring in these structures and their potential association with sports performance and/or injury predisposition will be explored. Overall, this study utilizes a comparative cross-sectional research design, where different groups are assessed regarding musculotendinous adaptations in the Achilles tendon and triceps surae through ultrasound-derived measures. The use of the VISA-A scale and the assessment of measure reliability will provide additional data on pain, function, and result reproducibility.

DETAILED DESCRIPTION:
Introduction: Triathlon is a growing sport worldwide, accompanied by a range of injuries primarily linked to the running component, with calcaneal tendinopathy standing out prominently due to the significant demands placed on this structure in both running and cycling. While numerous studies have assessed the architecture of triceps surae muscles and the Achilles tendon in athletes from various sports, exploring both positive and negative adaptations, as well as characteristics associated with improved performance or injury predisposition, there is a notable absence of research specifically investigating these tissues in triathletes. Understanding the architecture of the Achilles tendon and triceps surae muscles in this specific population is crucial for elucidating structural alterations related to performance and injurious changes in these structures. Ultrasound imaging emerges as the standard examination for evaluating these structures due to its quality, portability, and real-time information provision.

Objective: This study aims to identify musculotendinous adaptations in the Achilles tendon and muscles composing the triceps surae induced by triathlon training and competitions in both high-performance and low-performance athletes. These adaptations may be related to injury predisposition and could explain differences in sports performance between groups.

Methods: Twenty high-performance triathletes, twenty low-performance triathletes, and twenty physically active, healthy individuals of both genders will be screened through anamnesis to determine the research groups. Pain and function of the Achilles tendon will be measured using the VISA-A scale (Victorian Institute of Sport Achilles Assessment). The structure of the Achilles tendon and the muscular architecture of the triceps surae will be assessed through ultrasound imaging. The reliability of ultrasound measures will be determined by evaluating images of individuals using the intraclass correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

High and Low-Performance Triathlete Groups:

* Be a triathlete practicing the sport for more than one year.
* Have participated in and completed at least two triathlon events.
* Maintain regular training at least 4 times per week.
* Be between 17 and 52 years old.

Control Group:

* Be between 17 and 52 years old.
* Engage in regular physical activity (minimum 3 times per week).

Exclusion Criteria:

High and Low-Performance Triathlete Groups:

* Have any disease or injury limiting training and competitions at the time of assessment.
* Not have been training regularly in the last 2 weeks prior to assessment.
* Present acute inflammation, acute pain, or delayed onset muscle soreness on the assessment day.
* Use anabolic steroids.
* Have used steroidal anti-inflammatories in the last 4 weeks before assessment.
* Have used Fluoroquinolone antibiotics in the last 4 weeks before assessment, as they may alter collagen synthesis and induce tendinopathies (ALVES; MENDES; MARQUES, 2019).
* Engage in regular practice of another sport.

Control Group:

* Have any disease or injury limiting physical activity.
* Regularly engage in street running (run at least 20km per week).
* Present acute inflammation, acute pain, or delayed onset muscle soreness on the assessment day.
* Use anabolic steroids.
* Have used steroidal anti-inflammatories in the last 4 weeks before assessment.
* Have used Fluoroquinolone antibiotics in the last 6 months before assessment, as they may alter collagen synthesis and induce tendinopathies (ALVES; MENDES; MARQUES, 2019).
* Have regularly practiced street running at any point in life.

Ages: 17 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study participants must be triathletes, excluding the control group, of both genders, aged between 17 and 52 years, engaging in the sport for over a year, having completed at least two triathlon events, maintaining regular training at least four times a week, and having no limiting health conditions for training and event participation.
  It is important to note that all participants in the control group should engage in regular physical activity at least three times a week, excluding street running, and be aged between 17 and 52 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-07-16 (Estimated); Study Completion 2024-10-04 (Estimated)

PRIMARY OUTCOMES:
Morphological Properties: Tendon Length (TL). | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  To obtain the tendon length, the ultrasound probe will be placed longitudinally to the tendon. The most distal portion of the Achilles tendon inserted into the calcaneus bone will be visualized using ultrasound, and the corresponding point will be marked on the skin. Subsequently, the probe will be moved proximally until the visualization of the myotendinous junction (JMT) of the medial gastrocnemius muscle, and this point will also be marked on the skin. The distance between the two marked points on the skin will be measured using a tape measure, and this distance will be considered representative of the tendon length.
Evaluation of Achilles Tendon Shape (fusiform or parallel) | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  All Achilles tendons will be scanned in sagittal and axial planes, taking care to avoid anisotropy. The maximum thickness of the tendon (anterior to posterior) will be measured in sagittal and axial planes (between 3 and 6 cm above the tendon insertion in all cases), and this measurement has shown acceptable reliability (BRUSHØJ et al., 2006). As the Achilles tendon rotates medially from proximal to distal, the tendon thickness was measured very close but not always precisely in the sagittal plane.
  The ratio of the thickest portion to the enthesis will be calculated from static images saved at these measures. Tendons will be categorized as fusiform if this ratio is 4:1, indicating a 20% increase in thickness in the midportion compared to the enthesis (MALLIARAS et al., 2010).
Echogenicity of the Tendon (homogeneous and heterogeneous areas) | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  Echogenicity will be represented by a histogram on a grayscale with values ranging from 0 to 255 (0: black/no wave reflection; 255: white/total wave reflection). The measurement will be performed using the tracing method (VIEIRA et al., 2019), adopting the same region of interest (ROI) as described earlier for cross-sectional area calculation.
  Heterogeneous echogenicity will be defined as reduced echogenicity within the tendon seen in both sagittal and axial planes. Diffuse heterogeneous echogenicity will be defined when it presents focal hypoechoic regions (midportion and/or enthesis). Ten ROIs will be grouped based on echogenicity by a trained researcher (MALLIARAS et al., 2010).
Mechanical properties of the Achilles Tendon: Force | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The force (F) of the Achilles tendon will be calculated using equation 2 (Arya; Kulig, 2010; Geremia et al., 2018):
  F=ET/MA
  Calculation of force, where F is the force of the Achilles tendon, ET is the external torque, and MA is the moment arm of the Achilles tendon.
  The actual force of the Achilles tendon will be obtained by summing the torque value generated by the activation of the tibialis anterior muscle to the torque generated during plantar flexion, as per equation 3:
  F=TQp+TQat
  Calculation of Torque (TQ), where TQp is the torque generated by the plantar flexors, and TQat is the torque generated by the activation of the dorsal flexors during maximal isometric plantar flexion.
Mechanical properties of the Achilles Tendon: Stress | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The stress of the tendon will be calculated as the ratio of the force applied to the tendon to its cross-sectional area (CSA).
  Stress=F/CSA
  Calculation of stress, where F is the force of the Achilles tendon, and CSA is the cross-sectional area of the tendon.
Mechanical properties of the Achilles Tendon: Strain | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The strain in the tendon will be calculated using the change in the length of the TA in relation to the original length (ΔL/L0) during maximal voluntary contractions in the ramp protocol (ARYA; KULIG, 2010) and will be expressed as a percentage (GEREMIA et al., 2018).
  Strain=(Cf-Ci)/Ci.100
  Calculation of strain, where Cf is the final length of the Achilles tendon (length during contraction) and Ci is the initial length of the Achilles tendon (resting length). Stress and strain values will be obtained at 10% intervals of MVIC (from 0 to 100%) (GEREMIA et al., 2018).
Material Properties of the Achilles Tendon: Elastic Modulus | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  Elastic Modulus, also known as Young's Modulus, will be obtained by dividing stress by strain. Young's Modulus will be determined by the slope of the stress-strain curve (GEREMIA et al., 2018).
Muscle Thickness | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  For measuring muscle thickness, a line will be drawn in the thickest area of each muscle, between the superficial and deep aponeuroses, following the protocol of Arts et al., (2010).
Muscle Properties: Pennation Angle (PA) | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The pennation angle variable refers to the angle of the muscle fibers concerning the muscle's line of force. To measure it, the angle formed between a muscle fiber and the deep aponeurosis will be observed (LIMA; OLIVEIRA, 2013). The pennation angle (PA) will be calculated as the angle between the muscle fascicle and the deep aponeurosis.
Muscle Properties: Fascicle Length (FL) | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The Fascicle Length (FL) will be considered as the total length of the muscle fiber. However, as fascicles are too long to be measured from origin to insertion (i.e., the distance between aponeuroses and myotendinous junctions), the estimated length will be obtained using the formula of Blazevich et al. (2006), which uses muscle thickness, fascicle angle, and the angle between the superficial and deep fascia as variables. The best fascicle (i.e., the fascicle that can be seen in its entirety from its insertion into the deep aponeurosis to the superficial aponeurosis or to the end of the ultrasound probe's field of view) in each image will be used for FL and PA analysis. FL will be considered as the length of the fascicular path between the superficial and deep aponeuroses. When the ends of the fascicles are outside the ultrasound image, FL will be estimated as recommended in previous studies (ABELLANEDA; GUISSARD; DUCHATEAU, 2009; AVELA et al., 2004; FINNI, 2006).
Muscle Echogenicity | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The evaluation of echogenicity will be performed through grayscale analysis, where affected muscles appear whiter, i.e., hyperechoic, resulting from increased intramuscular fibrous and adipose tissue and zones of necrosis (PUTHUCHEARY et al., 2015). The echogenicity measurement region will be selected in each muscle to include the maximum possible muscle area without bone or surrounding fascia (PILLEN et al., 2006). With an 8-bit resolution, the images will result in values that can vary between 0 and 255 (0: black/no wave reflection; 255: white/total wave reflection), which will be performed by the tracing method (VIEIRA et al., 2019).
Assessment of Muscle Electrical Activation | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  The electrical activity of the medial gastrocnemius (GM) and tibialis anterior (TA) muscles will be assessed through electromyography (EMG), and the EMG system will be connected to the data acquisition system and synchronized with the isokinetic dynamometer, allowing the assessment of electrical activity during maximal isometric tests.
Muscle Torque Evaluation | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  Isometric torque assessment will be conducted through three maximal voluntary isometric contractions (MVICs) of plantar flexion and dorsiflexion at a joint position of 0° (foot surface perpendicular to the leg). Each isometric contraction will last for 5 seconds with a rest period of 2 minutes between contractions. The peak torque value for each contraction will be checked during data collection, and an additional maximal isometric test will be performed when the variation between the values obtained in the first three tests exceeds 10%. A standardized verbal stimulus will be given during all force tests to motivate participants to achieve their maximum strength. The highest peak torque values obtained during the isometric tests will be used for statistical analysis.
Evaluation of Muscle and Achilles Tendon Stiffness through 2D Shear Wave Elastography (SWE): | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  Muscle stiffness in triceps surae muscles will be assessed using Acuson Redwood Ultrasound System - Siemens®, USA. Musculoskeletal settings with 0-300 kilopascal (kPa) scales will be employed. B-mode ultrasound images, utilizing a linear transducer, will generate 30 circular Regions of Interest (ROIs) in different muscle regions. Shear wave velocity from these ROIs will determine muscle tissue stiffness. The average shear wave velocity across the three muscles will represent triceps surae stiffness. Achilles tendon stiffness will follow a similar process with nine manually chosen ROIs. Gel and a gel pad will ensure acoustic coupling. SWE assessments, by a consistent evaluator, will occur in a controlled temperature environment (23-25ºC). Three resting position images per tissue will be obtained, allowing a 10s delay for elastography map stabilization.

SECONDARY OUTCOMES:
Ankle pain and function | Assessment will occur during a single visit of the triathlete to the laboratory, specifically between the months of March to July 2024.
  To assess ankle pain and function in our research groups, we will use the Victorian Institute of Sport Achilles Assessment scale (VISA-A), developed by the Victorian Institute of Sport (Melbourne, Australia). It is a self-assessment tool, already translated into Brazilian Portuguese and validated. The scale consists of eight questions, with the first six on a visual analog scale and the last two on a categorical rating scale. The final questionnaire score ranges from 0 to 100, with 0 representing the worst condition and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: João LQ Durigan, PhD, Study Director — UnB

IPD SHARING:
Plan to Share IPD: No
The authors consider sharing the data depending on the situation.